CLINICAL TRIAL: NCT02718963
Title: Treatment of Dysphagia by Using a Synchronized Electrical Stimulation Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ju Seok Ryu, associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-1507/306-002
Record Dates: First submitted 2016-03-20; First posted 2016-03-24 (Estimated); Results first posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: Deglutition Disorders
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Experimental): * control group(N=10): who does not have dysphagia symptom
  * apply Synchronized Electrical Stimulation Device
    * before apply the synchronized electrical stimulation device, we will evaluate the high resolution manometry for evaluation of deglutition function
    * during apply the synchronized electrical stimulation device, we will evaluate the high resolution manometry for evaluation of deglutition function
  Interventions: Device: Synchronized Electrical Stimulation Device
- Experimental group (Experimental): * experimental group(N=10): who have dysphagia symptoms
  * apply Synchronized Electrical Stimulation Device
    * before apply the synchronized electrical stimulation device, we will evaluate the high resolution manometry for evaluation of deglutition function
    * during apply the synchronized electrical stimulation device, we will evaluate the high resolution manometry for evaluation of deglutition function
  Interventions: Device: Synchronized Electrical Stimulation Device

INTERVENTIONS:
Device: Synchronized Electrical Stimulation Device — electrical stimulation at muscles which related with deglutition

SUMMARY:
The purpose of this study is to determine the synchronized electrical stimulation device effective in the treatment of dysphagia.

DETAILED DESCRIPTION:
* Design: Prospective study
* Inclusion criteria of the patient group: who has a dysphagia symptom and confirmed by video-fluoroscopic swallowing study(N=10)
* Inclusion criteria of the control group: who does not have any dysphagia symptoms, and does not have any underlying disease(N=10)
* Setting: Hospital rehabilitation department
* Intervention: Participants are applied electrical stimulation by a "Synchronized Electrical Stimulation Device(SESD)"

ELIGIBILITY:
Inclusion Criteria:

* who have dysphagia symptoms and verified deglutition disorder by video fluoro swallowing study

Exclusion Criteria:

* who reject the checkup their deglutition function by high resolution manometry
* who reject apply "Synchronized Electrical Stimulator"

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2016-06-24 (Actual); Study Completion 2016-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jusuk Ryu, M.D. PhD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Department of Rehabilitation Medicine, Seoul National University Bundang Hospital, Seoul National University College of Medicine, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Park D, Suh JH, Kim H, Ryu JS. The Effect of Four-Channel Neuromuscular Electrical Stimulation on Swallowing Kinematics and Pressures: A Pilot Study. Am J Phys Med Rehabil. 2019 Dec;98(12):1051-1059. doi: 10.1097/PHM.0000000000001241. PMID 31180928
- [Derived] Lim J, Hyun SE, Kim H, Ryu JS. Residual effect of sequential 4-channel neuromuscular electrical stimulation evaluated by high-resolution manometry. Biomed Eng Online. 2024 Jul 25;23(1):70. doi: 10.1186/s12938-024-01269-1. PMID 39049019

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was no significant event in the study after participant enrollment
Groups:
- Control Group: * control group(N=10): who does not have dysphagia symptom
  * apply Synchronized Electrical Stimulation Device
    * before apply the synchronized electrical stimulation device, we will evaluate the high resolution manometry for evaluation of deglutition function
    * during apply the synchronized electrical stimulation device, we will evaluate the high resolution manometry for evaluation of deglutition function
  Synchronized Electrical Stimulation Device: electrical stimulation at muscles which related with deglutition
- Experimental Group: * experimental group(N=10): who have dysphagia symptoms
  * apply Synchronized Electrical Stimulation Device
    * before apply the synchronized electrical stimulation device, we will evaluate the high resolution manometry for evaluation of deglutition function
    * during apply the synchronized electrical stimulation device, we will evaluate the high resolution manometry for evaluation of deglutition function
  Synchronized Electrical Stimulation Device: electrical stimulation at muscles which related with deglutition
Period: Overall Study
Arm/Group | Control Group | Experimental Group
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Experimental Group | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (11.99) | 65.9 (13.06) | 58.75 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 6 | 8 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 10 | 10 | 20
Disease [Count of Participants; unit: Participants]
  Stroke | 0 | 4 | 4
  Brain tumor | 0 | 1 | 1
  Cerebral palsy | 0 | 1 | 1
  Guillain-Barre syndrome | 0 | 1 | 1
  Spinal cord injury | 0 | 1 | 1
  Unknown | 0 | 2 | 2
  Healthy | 10 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: Pressure and Timing Change of Velopharynx, Tongue Base, Low Pharynx and Upper Esophageal Sphincter.
Description: Maximal pressure, integral, rise time, and duration in the regions of VP and TB (the time interval over the VP and TB integral).
  The maximal pressure of low pharynx (LP) (C in supplementary 1), maximal pre-upper esophageal sphincter (UES) pressure (F in supplementary 1), maximal cricopharyngeus (CP) pressure (D in supplementary 1), minimal upper esophageal sphincter (UES) pressure, upper esophageal sphincter (UES) activity time (the interval between pre-upper esophageal sphincter (UES) peak and post-upper esophageal sphincter (UES) peak; G in supplementary 1), and nadir upper esophageal sphincter (UES) pressure duration in the region of upper esophageal sphincter (UES).
Time Frame: During the electrical stimulation and electrical stimulation effects of Velopharynx, tongue base, lower pharynx and upper esophageal sphincter
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 10 | 10
mmHg
  Control, pressure of VP, thin | 162.04 (39.67) | 129.66 (45.58)
  NMES, pressure of VP, thin | 200.90 (70.61) | 170.66 (77.10)
  Control, pressure of tongue base, thick | 81.59 (44.51) | 136.40 (27.20)
  NMES, pressure of tongue base, thick | 109.22 (54.36) | 151.26 (34.86)
Statistical Analysis 1: Comparison: Control Group vs Experimental Group; Wilcoxon signed rank test was used to compare the Videofluoroscopic swallowing study(VFSS) kinematic variables, VDS, PAS, and high resolution manometry (HRM) variables between the neuromuscular electrical stimulation session and the control session in swallowing thin fluid and thick fluid for healthy, dysphagic and whole participants. Mann-Whitney test was used to compare the differences of VFSS variables, VDS, PAS, and HRM variables between the healthy participants and dysphagic participants; Test type: Other; p < 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.05

ADVERSE EVENTS:
Time Frame: 3 days after finishing the examination.
Arm/Group | Control Group | Experimental Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
First, a small number of subjects were included. Second, the sequential 4-channel NMES was not directly compared with the 2-channel NMES. Third, some prospectively enrolled healthy participants in our study had asymptomatic penetration in VFSS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No